CLINICAL TRIAL: NCT02169843
Title: Influence of Small Doses Dexmedetomidine to the Elderly Patients' Emergence Agitation
Brief Title: Small Doses of Dexmedetomidine for Emergence Agitation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140523 Dexmedetomidine
Record Dates: First submitted 2014-05-26; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Emergence Agitation
Keywords: Dexmedetomidine,; agitation,; AFPS,; NRS,; mean arterial pressure; heart rate(HR)
MeSH Terms: conditions — Emergence Delirium; Psychomotor Agitation | interventions — Sevoflurane; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Sevoflurane & Dexmedetomidine (Experimental): inhale Sevoflurane + intravenous pumping Remifentanil 0.1µg/kg/min + intravenous inject cisatracurium besilate 0.08mg/kg in fixed time interval + finally add sufentanil 0.15µg/kg,and intravenous pumping Dexmedetomidine 0.2µg/kg/h.
  Interventions: Drug: Sevoflurane; Drug: Dexmedetomidine
- Sevoflurane & Placebo (Active Comparator): inhale Sevoflurane + intravenous pumping Remifentanil 0.1µg/kg/min + intravenous inject cisatracurium besilate 0.08mg/kg in fixed time interval + finally add sufentanil 0.15µg/kg,and intravenous pumping Placebo(for Dexmedetomidine )0.05ml/kg/h.
  Interventions: Drug: Sevoflurane; Drug: Placebo(for Dexmedetomidine)

INTERVENTIONS:
Drug: Sevoflurane — inhale Sevoflurane
  Other Names: Sevoflurome
Drug: Dexmedetomidine — intravenous pumping Dexmedetomidine 0.2µg/kg/h
  Other Names: Dexmedetomidine Hydrochloride Injection
  Arms: Sevoflurane & Dexmedetomidine
Drug: Placebo(for Dexmedetomidine) — normal saline mimic Dexmedetomidine, intravenous pumping 0.05ml/kg/h
  Other Names: normal saline
  Arms: Sevoflurane & Placebo

SUMMARY:
Dexmedetomidine Hydrochloride is a kind of high selectivity alpha 2 agonists adrenaline, can inhibit the activity of sympathetic nerve, and reduce the adverse effects of stress reaction in anesthesia recovery period.Literatures have been reported that Dex can reduce the rate of emergence agitation of children and adults,especially in elderly patients(>64 years) after using sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. obtain informed consent;
2. patients whose selective under general anesthesia colorectal cancer or esophageal cancer radical operation time > 2h;
3. the American society of anesthesiologists (ASA) class I-II;
4. age>64 years old;
5. BMI<28kg/㎡;

Exclusion Criteria:

1. systolic pressure≥180mm Hg or<90mm Hg, diastolic pressure≥110mm Hg or< 60mm Hg;
2. serious heart, brain, liver, kidney, lung, endocrine diseases or serious infections;
3. patients with difficult airway (such as Mallampati airway class III, airway abnormalities, etc.)
4. HR<50times/min
5. a history of mental illness or a long history of taking medicine of psychiatric drugs and chronic analgesics
6. a history of alcoholism
7. diseases of the neuromuscular
8. a tendency to malignant hyperthermia
9. allergy to test drugs or have other contraindications
10. participated in other clinical drug researches over the past 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
evaluation of agitation | the duration of PACU room stay,expect 30 minutes
  stay in the PACU room after operation,measure the score of Aono's four-point scale(AFPS) every two minutes.
evaluation of pain | the duration of PACU room stay,expect 30 minutes
  stay in the PACU room after operation,measure the score of numeric rating scale(NRS) every two minutes.
the amount of drugs | the duration of hospital stay,expect 5 weeks
  when stay in the hospital,measure the total doses of Nalbuphine and Fentanyl using
number of agitation | the duration of hospital stay,expect 5 weeks
  when stay in the hospital, measure the number of agitation.

SECONDARY OUTCOMES:
the mean arterial pressure | from the beginning of induction to skin closure, up to 1 hour
  measure the mean arterial pressure at 6 time points including after pump injection of Dexmedetomidine or normal saline 10 minutes, 20 minutes,30 minutes,before pulling out the endotracheal tube,at the time of pulling out the endotracheal tube,and after pulling out the endotracheal tube 5 minutes
heart rate | from the beginning of induction to skin closure, up to 1 hour
  measure the heart rate at 6 time points including after pump injection of Dexmedetomidine or normal saline 10 minutes, 20 minutes,30 minutes,before pulling out the endotracheal tube,at the time of pulling out the endotracheal tube,and after pulling out the endotracheal tube 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi’an, Shanxi, China